CLINICAL TRIAL: NCT00708006
Title: A Phase 1 Dose-Escalation Study to Evaluate the Safety and Tolerability of HGS1029 (AEG40826-2HCl) in Patients With Advanced Solid Tumors
Brief Title: A Study of HGS1029 (AEG40826-2HCl) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGS1029-C1078
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HGS1029
  Interventions: Drug: HGS1029

INTERVENTIONS:
Drug: HGS1029 — Escalating doses by IV (in the vein), on days 1, 8 and 15 of each 28-day cycle. Number of cycles: until disease progression or unacceptable toxicity
  Other Names: AEG40826•2HCl

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of HGS1029 in subjects with advanced solid tumors and to determine a phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced solid malignancy
* Life expectancy of at least 3 months
* Age 18 years or older
* Acceptable liver function
* Acceptable renal function
* Acceptable hematologic status

Exclusion Criteria:

* Received investigational (not yet approved by a regulatory authority)agent within 4 weeks before enrollment.
* Received non-investigational agent within 3 weeks before enrollment.
* Progressive CNS involvement including the need of corticosteroids
* Pregnant or breast-feeding women
* Active, uncontrolled bacterial, viral, or fungal infections within 2 weeks of Cycle 1 Day 1
* Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and dose-limiting toxicity of HGS1029 administered weekly X 3, repeated every 4 weeks | throughout the study

SECONDARY OUTCOMES:
Determination of pharmacokinetic profile; evaluation of biomarkers; evaluation of possible anti-tumor activity | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Gallant, B. Pharm.,Ph.D., Study Director — Human Genome Sciences Inc.
Locations (3):
- United States (3):
  - Stanford University Dept. of Medicine-Oncology, Stanford, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - The Sarah Cannon Research Institute, Nashville, Tennessee